CLINICAL TRIAL: NCT00651755
Title: Evaluation of Aprepitant's Effect on Drug Metabolism in Multi-Day Combination (CHOP/R-CHOP) Chemotherapy Regimen in Patients With Non-Hodgkin's Lymphoma
Brief Title: Aprepitant's Effect on Drug Metabolism in Multi-Day Combination (CHOP/R-CHOP) Chemotherapy Regimen in Lymphoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006-1033
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoma; Nausea; Cyclophosphamide; Cytoxan; Neosar; Doxorubicin; AD; Hydroxydaunomycin hydrochloride; Vincristine; Prednisone; Rituximab; Rituxan; Aprepitant; Emend; L754030; MK869; Drug Metabolism; CHOP; R-CHOP; NHL
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Nausea | interventions — Aprepitant; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Rituximab; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant + CHOP/R-CHOP (Experimental): Aprepitant 125 mg oral (PO) Day 1 of Cycle 1 followed by 80 mg PO Daily Days 2-3 with CHOP (steroid in CHOP) or R-CHOP plus Rituximab 375 mg/m^2 intravenous Day 1. CHOP or R-CHOP chemotherapy: (1) bolus or 48-hour infusion CHOP [cyclophosphamide 750 mg/m^2 IV Day 1, doxorubicin 25 mg/m^2/day IV given bolus or over 48 hours continuous infusion Days 1-2, vincristine 2 mg IV Day 1, prednisone PO 100 mg * 5 days]; or (2) Bolus or 48-hour infusion R-CHOP [Rituximab 375 mg/m^2 on Day 1 + CHOP as above]. [For patients receiving R-CHOP, CHOP may be administered starting on Day 2 at the discretion of the treating physician]
  Interventions: Drug: Aprepitant; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab
- Standard of Care (Control) + CHOP/R-CHOP (Experimental): Anti-emetics, Ondansetron 8 mg daily for 2 days, plus steroids in CHOP or R-CHOP regimen.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab; Drug: Ondansetron

INTERVENTIONS:
Drug: Aprepitant — 125 mg By Mouth (PO) On Day 1, followed by 80 mg PO Daily On Days 2-3.
  Other Names: Emend; L754030; MK869
  Arms: Aprepitant + CHOP/R-CHOP
Drug: Cyclophosphamide — 750 mg/m^2 By Vein On Day 1
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — 25 mg/m^2 By Vein Over 48 Hours On Days 1-2
  Other Names: AD; Hydroxydaunomycin hydrochloride
Drug: Vincristine — 2 mg By Vein On Day 1
Drug: Prednisone — 100 mg PO for 5 Days
Drug: Rituximab — 375 mg/m^2 By Vein On Day 1.
  Other Names: Rituxan
Drug: Ondansetron — 8 mg daily for 2 days
  Arms: Standard of Care (Control) + CHOP/R-CHOP

SUMMARY:
The goal of this clinical research study is to learn the effect of combining aprepitant with CHOP or R-CHOP in patients with Non-Hodgkin's Lymphoma (NHL) that is either newly diagnosed or has come back. Researchers also want to see if aprepitant can help to prevent nausea and/or vomiting that may be caused by chemotherapy treatment with CHOP or R-CHOP, in these patients. CHOP consists of four drugs - Cyclophosphamide (also called Cytoxan/Neosar), Doxorubicin (or Adriamycin), Vincristine (Oncovin) and Prednisolone while R-CHOP includes Rituximab and CHOP.

DETAILED DESCRIPTION:
The Study Drugs:

Aprepitant is designed to block the natural substance in the brain that causes nausea and vomiting. This may help to prevent and/or control nausea and vomiting caused by cancer chemotherapy treatment.

CHOP and R-CHOP are commonly used chemotherapy regimens for treating NHL.

In the blood, aprepitant may increase or decrease the drug levels of cyclophosphamide, vincristine, and/or prednisone (which are part of the CHOP and R-CHOP regimens), but this is not known for certain. This study is designed to help researchers learn the effect of combining aprepitant with CHOP and R-CHOP.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. There is an equal chance of being assigned to either group.

Standard Chemotherapy Administration:

Both CHOP and R-CHOP typically have 21-day "cycles" but can vary from every 14 to 28 days. You will receive CHOP or R-CHOP according to the schedule prescribed by your doctor. You will also receive standard medications for preventing nausea and vomiting. You will sign a separate consent form that will describe these treatments in detail, along with their risks.

Aprepitant Administration:

Aprepitant is taken by mouth, with or without food.

Group 1 will take aprepitant on Days 1, 2, and 3 of Study Cycle 1 only. Group 2 will take aprepitant on Days 1, 2, and 3 of Study Cycle 2 only.

Study Diary:

Prior to each study cycle, you will be given a study diary to use throughout the study. Once a day, you will record any side effects you may have experienced. You should bring your study diary to every study visit so the study staff can review it.

Study Visits:

Prior to each study cycle, you will have a study visit with the following tests/procedures performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of vital signs and weight.
* You will have a performance status evaluation.
* You will fill out the same questionnaire you did at screening, about any nausea and vomiting you may be experiencing.
* You will be asked about any other medications you may be taking. Be sure to tell the study doctor about all medications (including vitamins, herbal products, and nutritional supplements), because some medications/substances will cause side effects when taken at the same time as aprepitant.
* The study staff will review your study diary.

Pharmacokinetic Testing:

You will have additional blood samples drawn for pharmacokinetic (PK) testing of cyclophosphamide, vincristine, and prednisone levels. PK testing measures the amount of the drug in the body at different time points. These PK blood draws will be about 2 tablespoons each.

On Days 1 and 2 of Study Cycles 1 and 2, blood will be drawn for PK testing at the following times: before taking prednisone, 30 minutes after the start of the cyclophosphamide infusion, and at 60 minutes, 75 minutes, 90 minutes, and 2, 4, 6, 8, and 24 hours after the start of the cyclophosphamide infusion.

Other Blood Tests:

At least twice a week during Study Cycles 1 and 2, blood (about 1 teaspoon) will be drawn for routine tests.

Aprepitant may increase the blood sugar during the first few days the drug is taken. Because of this, on Day 1 of Study Cycle 1, you will be given a glucometer (a machine to check your blood sugar). You will use the glucometer at home during the study (or in the hospital if you are admitted there for chemotherapy). You will be given instructions on how to use it, and what to be looking for. On Days 1-6 of Study Cycle 1, you will give yourself a "fingerstick" blood sugar test once a day (before breakfast). You will take a "fingerstick" blood sugar test before you receive each dose of aprepitant.

Length of Study:

You may receive up to 2 cycles of chemotherapy, including 1 cycle of aprepitant. If intolerable side effects occur or the disease gets worse, you will be taken off study early.

End-of-Study Visit:

At 30 days after your last dose of aprepitant, you will return for an end-of-study visit. At this visit, you will have the same tests/procedures performed that you did at the other study visits. You will return the glucometer to the study staff.

This is an investigational study. The CHOP and R-CHOP regimens are commercially available and FDA approved for use in NHL.

Aprepitant is commercially available and FDA approved (when used in combination with other nausea medication, such as ondansetron) for the prevention of nausea and vomiting that may be caused by chemotherapy. However, this study is considered experimental because researchers want to find out how aprepitant may affect the drug levels of cyclophosphamide, vincristine, and prednisone in the blood. (Cyclophosphamide, vincristine, and prednisone are part of the CHOP and R-CHOP regimens.) The use of aprepitant is authorized for this experimental purpose.

Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or relapsed lymphoid malignancy.
2. Patients receiving either:(1) Bolus or 48-hr infusion CHOP (cyclophosphamide 750 mg/m^2 IV Day 1, doxorubicin 25 mg/m^2/day IV given as bolus infusion or over 48 hours continuous infusion Days 1-2, vincristine 2 mg IV Day 1, prednisone PO 100 mg * 5 days) OR (2) Bolus or 48-hr infusion R-CHOP (Rituximab 375mg/m^2 on Day 1+ CHOP as above). (For patients receiving R-CHOP, CHOP may be administered starting on Day 2 at the discretion of the treating physician
3. Age >/= to 18 years
4. Adequate organ function defined as serum total bilirubin </= 1.2 mg/dL, serum aspartate aminotransferase or serum glutamate oxaloacetate transaminase (SGOT) </= 60 IU/L, creatinine < 1.5 mg/dL.

Exclusion Criteria:

1. Evidence of neoplastic central nervous system disease
2. Patients who are unable to take oral medication (e.g. due to tumor obstruction)
3. History of Diabetes Mellitus (Diabetes as defined by established diagnosis of diabetes currently receiving medications for the diabetes management and/or a fasting blood glucose of >/= 126 mg/dL.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 14, 2008 to May 3, 2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 23 participants who enrolled, three (3) withdrew prior to group assignment and were excluded from the trial.
Groups:
- First Aprepitant Cycle 1 Then No Aprepitant Cycle 2: First Aprepitant with CHOP or R-CHOP (CHOP plus Rituximab 375 mg/m^2 intravenous Day 1) then No Aprepitant in Cycle 2.
  Aprepitant 125 mg oral (PO) Day 1 of Cycle 1 followed by 80 mg PO Daily Days 2-3 with CHOP (steroid in CHOP) or R-CHOP plus Rituximab 375 mg/m^2 intravenous Day 1. CHOP or R-CHOP chemotherapy: (1) bolus or 48-hour infusion CHOP [cyclophosphamide 750 mg/m^2 IV Day 1, doxorubicin 25 mg/m^2/day IV given bolus or over 48 hours continuous infusion Days 1-2, vincristine 2 mg IV Day 1, prednisone PO 100 mg * 5 days]; or (2) Bolus or 48-hour infusion R-CHOP [Rituximab 375 mg/m^2 on Day 1 + CHOP as above].
- First No Aprepritant Cycle 1, Then Aprepitant Cycle 2: First No Aprepitant in Cycle 1, then Aprepitant 125 mg oral (PO) Day 1 of Cycle 2 followed by 80 mg PO Daily Days 2-3 with CHOP (steroid in CHOP) or R-CHOP plus Rituximab 375 mg/m^2 intravenous Day 1. CHOP or R-CHOP chemotherapy: (1) bolus or 48-hour infusion CHOP [cyclophosphamide 750 mg/m^2 IV Day 1, doxorubicin 25 mg/m^2/day IV given bolus or over 48 hours continuous infusion Days 1-2, vincristine 2 mg IV Day 1, prednisone PO 100 mg * 5 days]; or (2) Bolus or 48-hour infusion R-CHOP [Rituximab 375 mg/m^2 on Day 1 + CHOP as above].
Period: Cycle 1 (First 21 Days)
Arm/Group | First Aprepitant Cycle 1 Then No Aprepitant Cycle 2 | First No Aprepritant Cycle 1, Then Aprepitant Cycle 2
Started | 11 | 9
Completed | 10 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Cycle 2 (Second 21 Days)
Arm/Group | First Aprepitant Cycle 1 Then No Aprepitant Cycle 2 | First No Aprepritant Cycle 1, Then Aprepitant Cycle 2
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Not Evaluable | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Participants randomized to Aprepitant or control (Standard of Care) in Cycle 1 crossover for different treatment in Cycle 2.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age Continuous [Median (Full Range); unit: years] | 58 [22 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Area Under Curve (AUC) of Analyte, Cyclophosphamide (CP), in Aprepitant Treatment and Control Group
Description: Pharmacokinetic (PK) blood sampling to determine the geometric mean AUC of Cyclophosphamide (CP) during & post chemotherapy infusion, baseline, at 30, 60, 75, 90 minutes, and 2 , 4, 6, 8, and 24 hours from start of cyclophosphamide infusion. The absence of PK drug interactions was determined if the 90% Confidence Intervals (CI) of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25. Measurements reported as concentrate times the time, i.e. micrograms (ug)/milliliters (mL) times hour (hr).
Time Frame: Time points over 24 hours of cyclophosphamide infusion for both cycles (21 day cycle)
Population: There were 18 participants eligible for PK analysis, one was excluded from the final analysis due to data issues.
Measure: Geometric Mean (90% Confidence Interval); unit: ug/mL*hr
Groups:
- Aprepitant: Crossover study where participants received Aprepitant 125 mg oral (PO) Day 1 in Cycle 1 and received standard of care in Cycle 2. Or participants received no Aprepitant in Cycle 1, Aprepitant 125 mg oral (PO) Day 1 in Cycle 2.
- Control Group: Crossover study where participants received Standard of care in cycle 1 or cycle 2.
Arm/Group | Aprepitant | Control Group
Number analyzed (Participants) | 17 | 17
ug/mL*hr | 300 [276 to 326] | 250 [227 to 277]
Statistical Analysis 1: Comparison: Aprepitant vs Control Group; Test type: Non-Inferiority or Equivalence — The absence of pharmacokinetic drug interactions can be determined if the 90% CI of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25; 90% CI; Ratio Geometric Mean AUC = 1.20, 90% CI 2-sided [1.08 to 1.33] — Ratio Geometric Mean AUC (Area Under Curve) of Analyte,CP, between Aprepitant treatment to control Group

2. Primary Outcome: Geometric Mean Area Under Curve (AUC) of Analyte, 2-dechloro-cyclophosphamide(2-deCI-CP), in Aprepitant Treatment and Control Group
Description: Pharmacokinetic (PK) blood sampling to determine the geometric mean AUC of 2-deCI-CP, during & post chemotherapy infusion, baseline, at 30, 60, 75, 90 minutes, and 2 , 4, 6, 8, and 24 hours from start of cyclophosphamide infusion. The absence of PK drug interactions was determined if the 90% Confidence Intervals (CI) of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25. Measurements reported as concentrate times the time, i.e. micrograms (ug)/milliliters (mL) times hour (hr).
Time Frame: Time points over 24 hours of cyclophosphamide infusion for both cycles (21 day cycle)
Population: There were 18 participants eligible for PK analysis, one was excluded from the final analysis due to data issues.
Measure: Geometric Mean (90% Confidence Interval); unit: ug/mL*hr
Groups:
- Control: Crossover study where participants received Standard of care in cycle 1 or cycle 2.
Arm/Group | Aprepitant | Control
Number analyzed (Participants) | 17 | 17
ug/mL*hr | 4.5 [3.7 to 5.4] | 6.0 [4.8 to 7.5]
Statistical Analysis 1: Comparison: Aprepitant vs Control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; equivalence analysis; ratio Geometric mean AUC = 0.75, 95% CI 2-sided [0.65 to 0.86], Standard Deviation 0.29 — The geometric mean AUC ratio is the ratio of geometric mean AUC between aprepitant treatment and the control group

3. Primary Outcome: Geometric Mean Area Under Curve (AUC) of Analyte, 4-hydroxy-cyclophosphamide (4-OH-CP), in Aprepitant Treatment and Control Group
Description: Pharmacokinetic (PK) blood sampling to determine the geometric mean AUC of 4-hydroxy-cyclophosphamide (4-OH-CP), during & post chemotherapy infusion, baseline, at 30, 60, 75, 90 minutes, and 2 , 4, 6, 8, and 24 hours from start of cyclophosphamide infusion. The absence of PK drug interactions was determined if the 90% Confidence Intervals (CI) of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25. Measurements reported as concentrate times the time, i.e. micrograms (ug)/milliliters (mL) times hour (hr).
Time Frame: Time points over 24 hours of cyclophosphamide infusion for both cycles (21 day cycle)
Population: There were 18 participants eligible for PK analysis, one was excluded from the final analysis due to data issues.
Measure: Geometric Mean (90% Confidence Interval); unit: ug/mL*hr
Arm/Group | Aprepitant | Control
Number analyzed (Participants) | 17 | 17
ug/mL*hr | 3.9 [3.4 to 4.4] | 4.0 [3.4 to 4.7]
Statistical Analysis 1: Comparison: Aprepitant vs Control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; equivalence analysis; The geometric mean AUC ratio is the ratio of geometric mean AUC between aprepitant treatment to the control group; Ratio Geometric Mean AUC = 0.97, 90% CI 2-sided [0.83 to 1.13], Standard Deviation 0.35 — Ratio Geometric Mean AUC of Analyte, 4-OHCP, between Aprepitant treatment to control Group

4. Primary Outcome: Geometric Mean Area Under Curve (AUC) of Analyte, Vincristine (VC), in Aprepitant Treatment and Control Group
Description: Pharmacokinetic (PK) blood sampling to determine the geometric mean AUC of VC, during & post chemotherapy infusion, baseline, at 30, 60, 75, 90 minutes, and 2 , 4, 6, 8, and 24 hours from start of cyclophosphamide infusion. The absence of PK drug interactions was determined if the 90% Confidence Intervals (CI) of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25. Measurements reported as concentrate times the time, i.e. nanograms (ng)/milliliters (mL) times hour (hr).
Time Frame: Time points over 24 hours of cyclophosphamide infusion for both cycles (21 day cycle)
Population: There were 18 patients eligible for PK analysis, two participants were excluded from the analysis due to data issues.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL*hr
Arm/Group | Aprepitant | Control
Number analyzed (Participants) | 16 | 16
ng/mL*hr | 41 [34 to 49] | 39 [34 to 46]
Statistical Analysis 1: Comparison: Aprepitant vs Control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; equivalence analysis; Ratio Geometric Mean AUC = 1.04, 90% CI 2-sided [0.82 to 1.33], Standard Deviation 0.68 — Ratio Geometric Mean AUC (Area Under Curve) of Analyte, VC, Between Aprepitant treatment to control Group

5. Primary Outcome: Geometric Mean Area Under Curve (AUC) of Analyte,Prednisone (PR), in Aprepitant Treatment and Control Group
Description: Pharmacokinetic (PK) blood sampling to determine the geometric mean AUC of PR, during & post chemotherapy infusion, baseline, at 30, 60, 75, 90 minutes, and 2 , 4, 6, 8, and 24 hours from start of cyclophosphamide infusion. The absence of PK drug interactions was determined if the 90% Confidence Intervals (CI) of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25. Measurements reported as concentrate times the time, i.e. nanograms (ng)/milliliters (mL) times hour (hr).
Time Frame: Time points over 8 hours of cyclophosphamide infusion for both cycles (21 day cycle)
Population: Per protocol, 18 participants were eligible for PK analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL*hr
Arm/Group | Aprepitant | Control
Number analyzed (Participants) | 18 | 18
ng/mL*hr | 287 [262 to 315] | 265 [243 to 289]
Statistical Analysis 1: Comparison: Aprepitant vs Control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; equivalence analysis; Ratio Geometric Mean AUC = 1.08, 90% CI [1.02 to 1.15], Standard Deviation 0.17 — The geometric mean AUC ratio is the ratio of geometric mean AUC between aprepitant treatment and the control group

6. Primary Outcome: Geometric Mean Area Under Curve (AUC) of Analyte, Prednisolone (PL), in Aprepitant Treatment and Control Group
Description: Pharmacokinetic (PK) blood sampling to determine the geometric mean AUC of PL, during & post chemotherapy infusion, baseline, at 30, 60, 75, 90 minutes, and 2 , 4, 6, 8, and 24 hours from start of cyclophosphamide infusion. The absence of PK drug interactions was determined if the 90% Confidence Intervals (CI) of the geometric mean AUC ratio between 2 groups is within 0.80 to 1.25. Measurements reported as concentrate times the time, i.e. nanograms (ng)/milliliters (mL) times hour (hr).
Time Frame: Time points over 8 hours of cyclophosphamide infusion for both cycles (21 day cycle)
Population: Per protocol, 18 participants were eligible for PK analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL*hr
Arm/Group | Aprepitant | Control
Number analyzed (Participants) | 18 | 18
ng/mL*hr | 4416 [4027 to 4842] | 3817 [3324 to 4382]
Statistical Analysis 1: Comparison: Aprepitant vs Control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; equivalence analysis; Ratio Geometric Mean AUC = 1.16, 90% CI 2-sided [1.01 to 1.32], Standard Deviation 0.47 — Ratio Geometric Mean AUC (Area Under Curve) of Analyte,PL, Between Aprepitant treatment to control Group

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Groups:
- Aprepitant: Aprepitant 125 mg oral (PO) Day 1 (Cycle 1 or Cycle 2) to include treated study population.
- Control: Standard of Care
Arm/Group | Aprepitant | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=20) | Control (N=20)
Headache (General disorders) | 6 (6) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No